CLINICAL TRIAL: NCT02350062
Title: Comparison of Two Neuromuscular Monitors
Acronym: NMT-STIMPOD
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 13-183
Record Dates: First submitted 2014-11-27; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Neuromuscular Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Different neuromuscular monitors may be available in the same care structure. Two different monitors are available in the investigators' institution in the operative room and the recovery room. However, these two monitors have not been compared and may not be interchangeable. Starting the monitoring with one device and continuing with another device may be inaccurate and may lead to inadequate medical decisions. The investigators therefore conducted this observational study to compare the two devices available in our institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vascular surgery under general anesthesia and requiring neuromuscular blockade for intubation or surgery

Exclusion Criteria:

* Pregnancy or feeding
* Any pathology or medication that may impair neuromuscular conduction or muscular response of the ulnar nerve stimulation
* American Society of Anesthesiology [4] physical status
* Allergy or contraindication of neuromuscular blocking agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing vascular surgery under general anesthesia and requiring neuromuscular blockade for intubation or surgery
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Time to recover T4/T1 > 90% | Time between muscle relaxant injection and: intubation; recovery of 4 responses on the train of four (TOF); recovery of T4/T1 >40%; recovery of T4/T1>90% average 2 hours
  After muscle relaxant injection, we measure the time needed for the muscular response to disappear and to completely recover during the operation (which takes in average 2 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Georges Daccache, M.D, Principal Investigator — University Hospital, Caen